CLINICAL TRIAL: NCT06635460
Title: The Impact of Motivational Interviewing and Social Media-Based Patient Monitoring on Metabolic Control and Self-Efficacy in Adolescents With Type 1 Diabetes: A Randomized Controlled Trial
Brief Title: Motivational Interviewing and WhatsApp-Based Monitoring for Metabolic Control and Self-Efficacy in Adolescents With T1DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Büşra Kütük, Assistant Researcher, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 26.03.2024/03-27
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Type 1 Diabetes Mellitus (T1DM); Motivational Interviewing; Metabolic Control
Keywords: Type 1 diabetes mellitus; adolescent; motivational interviewing; social media-based monitoring; metabolic control; Self efficacy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: In the randomization scheme of the study, stratified and blocked randomization methods will be utilized. Age and gender variables will be used for the stratification of adolescents. Blocks will be formed as follows: for the age variable, "12-14 years" and "15-18 years" will be the categories, while for the gender variable, the categories will be "female" and "male." An online tool for generating blocked randomization lists will be employed. To achieve the calculated sample size for the study, each stratum will be repeated 7 times (2X2X7), resulting in a total inclusion of 56 adolescents, with each group comprising 28 participants.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Adolescents in this group will be followed up according to the routine follow-up program of pediatric endocrinology. Adolescents in the control group will not receive any intervention from the researcher during the study.
- Intervention Group (Experimental): Adolescents in this group will receive motivational interviewing and WhatsApp-based follow-up. Adolescents will be followed for 6 months. Online motivational interviewing sessions will occur once during the first 4 weeks. Meetings will then continue at 15-day intervals in the form of online motivational interview meetings and WhatsApp chats, respectively. Follow-up WhatsApp meetings will be held every 15 days for the next 3 months. The meetings will be conducted according to the "Intervention Group Meeting Content" prepared in accordance with the literature and expert opinion. The duration of the motivational meetings will be limited to 30-45 minutes in accordance with the literature. Blood glucose results, the lowest and highest values, and the reasons will be included in the content of patient follow-up, which will be conducted at intervals on the WhatsApp platform. Although the duration of written dialogues will vary among adolescents, it will be limited to an average of 2-10 min.
  Interventions: Other: Motivational interviewing; Other: Social media-based patient monitoring

INTERVENTIONS:
Other: Motivational interviewing — This programme has been developed from the literature and structured according to expert opinion. It will consist of a total of 8 online sessions. The duration of the motivational interviewing sessions will be limited to 30-45 minutes, in line with the literature.
  Arms: Intervention Group
Other: Social media-based patient monitoring — Blood glucose results, lowest and highest values, and reasons will be included in the content of the patient follow-up, which will be conducted at intervals on the WhatsApp platform. There will be a total of 10 follow-ups. Although the duration of the written dialog will vary among adolescents, it will be limited to an average of 2-10 minutes.
  Arms: Intervention Group

SUMMARY:
This clinical study aims to determine the effects of motivational interviewing and social media-based patient monitoring on metabolic control and self-efficacy in adolescents with Type 1 diabetes. Additionally, the study will assess the adolescents' attitudes toward their disease, quality of life, and perceived levels of social support. The primary research questions are as follows:

For adolescents with Type 1 diabetes who receive motivational interviewing and social media-based monitoring:

How do their attitudes toward their disease compare to those in the control group? How do their perceived levels of social support compare to those in the control group? How do their self-efficacy levels compare to those in the control group? How does their quality of life compare to that of the control group? How do their HbA1c levels compare to those in the control group?

DETAILED DESCRIPTION:
One of the most common chronic diseases in adolescence is type 1 diabetes mellitus (T1DM). T1DM is one of the most common endocrine diseases of childhood and requires lifelong management. To minimize the impact of T1DM on adolescents, metabolic control should be ensured, self-efficacy should be gained, quality of life should be improved, and anxiety should be reduced.

Because the epidemiology, pathophysiology, developmental status, and response to diabetes treatment are different in adolescents than in adults with diabetes, the care of adolescents should be different from that of adults. This population should be managed by a multidisciplinary team trained in pediatric diabetes management and sensitive to the difficulties of adolescents with T1DM. The diabetes nurse in this team is responsible for providing diabetes self-management education and support, medical nutrition therapy, and psychosocial support during and regularly after diagnosis. Interventions should focus on empowering adolescents to better manage their disease. Educational programs should include approaches such as teaching specific diabetes management skills and developing independence in these tasks (e.g., carbohydrate counting, blood glucose monitoring) and promoting autonomy and motivation.

Motivational interviewing techniques can be used to elicit behavior change by helping patients identify and resolve ambivalent feelings. Motivational interviewing is defined as a collaborative approach that elicits intrinsic motivation and strengthens commitment to behavior change goals. Motivating patients makes them feel ready to change their behavior and ensures that interventions to improve diabetes management are effective. Recent studies have shown that motivational interviewing also has a positive impact on diabetes self-management.

Today, social media is a valuable tool for people with diabetes to improve their self-management skills. Lifestyle changes such as diet and exercise, blood glucose monitoring, online education, peer support, and real-time interaction between patients and healthcare professionals can all be facilitated through social media. Therefore, it is recommended that healthcare professionals use social media-based applications to improve diabetes self-management skills and thereby improve glycemic control. This study will determine the effect of motivational interviewing and social media-based patient monitoring on metabolic control and self-efficacy in adolescents with type 1 diabetes. It will also determine the attitudes of adolescents with T1DM toward their own disease, quality of life, and perceived level of social support.

ELIGIBILITY:
Inclusion criteria:

* 13-18 years old,
* Diagnosed with type 1 DM at least 6 months ago,
* HbA1C level >7.0,
* 3-monthly outpatient visits,
* Completed basic type 1 DM education and scored high (≥15 points) on the Type 1 Diabetes Knowledge Assessment Form,
* A WhatsApp user with a smart phone and internet access,
* Adolescents who can speak and understand Turkish.

Exclusion criteria:

* Using an insulin pump,
* Having a chronic disease other than diabetes,
* Cognitive, intellectual, hearing, vision, or speech disabilities

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c test | At the beginning of the study (pre-test), 3 months after the pre-test, 6 months after the pre-test
  Participants will undergo HbA1c testing every 3 months throughout the study. These tests will serve as a long-term indicator of blood sugar control and one of the primary outcome measures of the study.
Diabetes Management Self-Efficacy Scale | At the beginning of the study (pre-test), 6 months after the pre-test
  The scale is used to assess the educational needs of adolescents or to evaluate the effectiveness of diabetes education programmes. The scale has 26 items. It has a Likert-type rating from 1 (strongly agree) to 5 (strongly disagree). The scale score is calculated by dividing the total self-efficacy score by the number of items to show the strength of perceived self-efficacy for different levels of performance. The minimum total score is 26 and the maximum is 130. A higher score indicates lower self-efficacy.

SECONDARY OUTCOMES:
Pediatric Quality of Life Inventory (PedsQL) 3.0 Diabetes Module | At the beginning of the study (pre-test), 6 months after the pre-test
  The 28-item multidimensional PedsQL 3.0 Diabetes Module included five subscales, which are diabetes symptoms (11 items), treatment barriers (4 items), treatment adherence (7 items), worry (3 items), and communication (3 items). The format, instructions, Likert type response scale, and the scoring method are identical to the PedsQL, with higher scores indicating fewer symptoms or problems.
Child Attitude Toward Illness Scale (CATIS) | At the beginning of the study (pre-test), 6 months after the pre-test
  The scale was developed to measure the attitudes of children with chronic illnesses towards their illness. The thirteen-item scale is scored as follows: 9 items were scored as 'very often, often, sometimes, not often, never' and 4 items were scored as 'very good, somewhat good, not sure, somewhat bad, very bad'. The scores for the 13 items were summed and divided by 13. The average score is between 1 and 5. Scores of 1 and 2 indicate a negative attitude, 3 a neutral attitude and 4 and 5 a positive attitude.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Kütük, Study Chair — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: July through December of 2026
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.

REFERENCES:
- [Background] Powell PW, Hilliard ME, Anderson BJ. Motivational interviewing to promote adherence behaviors in pediatric type 1 diabetes. Curr Diab Rep. 2014 Oct;14(10):531. doi: 10.1007/s11892-014-0531-z. PMID 25142716
- [Background] Guo J, Yang J, Wiley J, Ou X, Zhou Z, Whittemore R. Perceived stress and self-efficacy are associated with diabetes self-management among adolescents with type 1 diabetes: A moderated mediation analysis. J Adv Nurs. 2019 Dec;75(12):3544-3553. doi: 10.1111/jan.14179. Epub 2019 Oct 6. PMID 31441523
- [Background] American Diabetes Association. 13. Children and Adolescents: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S180-S199. doi: 10.2337/dc21-S013. PMID 33298424
- [Background] Al Ksir K, Wood DL, Hasni Y, Sahli J, Quinn M, Ghardallou M. Motivational interviewing to improve self-management in youth with type 1 diabetes: A randomized clinical trial. J Pediatr Nurs. 2022 Sep-Oct;66:e116-e121. doi: 10.1016/j.pedn.2022.05.001. Epub 2022 May 12. PMID 35568602
- [Background] Bakir E, Cavusoglu H, Mengen E. Effects of the Information-Motivation-Behavioral Skills Model on Metabolic Control of Adolescents with Type 1 Diabetes in Turkey: Randomized Controlled Study. J Pediatr Nurs. 2021 May-Jun;58:e19-e27. doi: 10.1016/j.pedn.2020.11.019. Epub 2020 Dec 25. PMID 33371976